CLINICAL TRIAL: NCT01241344
Title: A Randomized, Placebo-controlled, Multi-site Phase 2 Study Evaluating the Safety and Efficacy of Preemptive Treatment With CMX001 for the Prevention of Adenovirus Disease Following Hematopoietic Stem Cell Transplantation
Brief Title: Phase 2 Study to Evaluate Brincidofovir for the Prevention of Adenovirus Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMX001-202
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Results first posted 2021-07-16 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Adenovirus Disease
Keywords: AdV; Hematopoeitic Stem Cell Transplant; HSCT
MeSH Terms: interventions — brincidofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brincidofovir (Active Comparator): * Adult subjects: 200mg BCV administered as 50mg tablets taken orally either once weekly (QW; 4 tablets) or twice weekly (BIW; 2 tablets).
  * Pediatric subjects: 4mg/kg BCV (not to exceed a total single dose of 200mg) administered using a 10 mg/mL liquid formulation taken orally either QW (as 4 mg/kg) or BIW (as 2 mg/kg).
  Interventions: Drug: Brincidofovir
- Placebo (Placebo Comparator): * Adult subjects: Matching placebo tablets taken orally either once weekly (QW; 4 tablets) or twice weekly (BIW; 2 tablets).
  * Pediatric subjects: Matching liquid placebo taken orally either QW (as 4 mg/kg) or BIW (as 2 mg/kg).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Brincidofovir — * Adult subjects: 200mg BCV administered as 50mg tablets taken orally either once weekly (QW; 4 tablets) or twice weekly (BIW; 2 tablets).
  * Pediatric subjects: 4mg/kg BCV (not to exceed a total single dose of 200mg) administered using a 10 mg/mL liquid formulation taken orally either QW (as 4 mg/kg) or BIW (as 2 mg/kg).
  Other Names: BCV; CMX001
  Arms: Brincidofovir
Other: Placebo — Adult subjects: Matching placebo tablets taken orally either once weekly (QW; 4 tablets) or twice weekly (BIW; 2 tablets).
  • Pediatric subjects: Matching liquid placebo taken orally either QW (as 4 mg/kg) or BIW (as 2 mg/kg).
  Arms: Placebo

SUMMARY:
This study was designed to assess the safety and efficacy of preemptive treatment with oral brincidofovir (BCV), as compared to placebo, for the prevention of adenovirus (AdV) disease in recipients of hematopoietic stem cell transplantation (HCT) with asymptomatic AdV viremia.

DETAILED DESCRIPTION:
This was a Phase 2, randomized, multicenter, placebo-controlled study for pediatric and adult subjects who had undergone hematopoietic stem cell transplantation (HCT) and who had been identified as having asymptomatic adenovirus (AdV) viremia [i.e., had detectable AdV DNA in plasma based on polymerase chain reaction testing performed at the local laboratory with no AdV disease symptoms]. The primary objectives of the study were to assess the safety and tolerability of oral brincidofovir (BCV), and to estimate the treatment failure rate based on an efficacy endpoint with 2 different dosing regimens of oral BCV versus placebo.

ELIGIBILITY:
Inclusion Criteria

For inclusion into the study, subjects were required to fulfill all of the following criteria:

1. Were males or female aged ≥3 months to ≤75 years.
2. Received an allogeneic hematopoietic stem cell transplant (HCT).
3. Had positive serum adenovirus (AdV) PCR (>100 copies/mL) as measured by the central laboratory (unless the subject developed AdV disease while participating in the prescreening activities and after concurrence from the Chimerix medical monitor or designee).
4. Was on dialysis during treatment if he/she had an estimated glomerular filtration rate (eGFR) ≤30 mL/minute.
5. Subject or guardian(s) were willing to comply with the protocol.
6. Subject or guardian(s) were willing and able to understand the informed consent/assent.
7. Female subjects of child-bearing potential must have had a negative pregnancy test and must have agreed to use 2 acceptable methods of birth control throughout the study with at least 1 being a barrier method. Sexually active males of procreation potential must have been able and willing to se a reliable and medically approved contraceptive method throughout the study. At least 1 barrier method of contraception must have been used.

Exclusion Criteria

Subjects meeting any of the following exclusion criteria were excluded from participation in the study:

1. Had possible, probable, or definitive AdV disease (unless the subject developed probable or definitive AdV disease while participating in prescreening activities and after concurrence from he Chimerix medical monitor or designee).
2. Had suspected gut graft versus host disease that was not biopsy-proven (subjects with a biopsy performed were included in the study).
3. Had an eGFR ≤30 mL/minute and was not currently on dialysis.
4. Had an alanine aminotransferase or aspartate aminotransferase >5 x the upper limit of normal (ULN), total bilirubin ≥2 x the ULN, or conjugated (direct) bilirubin ≥1.5 x the ULN.
5. Had a condition that prevented oral dosing of study drug.
6. Was HIV antibody positive, based upon available medical records.
7. Had ocular hypotony, uveitis, or retinitis or any other intraocular pathology that would have predisposed the subject to 1 of these conditions.
8. Had participated in another clinical study of an investigational drug/biologic or was exposed to an investigational drug/biologic within 30 days of enrollment without the prior written approval of the Chimerix medical monitor or designee. For subjects who were participating in any clinical study involving non-investigational drugs and/or biologics, the investigator must have obtained approval from the Chimerix medical monitor or designee prior to enrolling the subject.
9. Was pregnant or breast-feeding or intended to conceive during the course of the study, including the follow-up period after drug discontinuation.
10. Had known immunologic hypersensitivity to cidofovir (CDV) or brincidofovir (BCV) drug or any of its excipients.
11. Had a history of illicit drug use or alcohol abuse within the previous 6 months.
12. Had any medical condition that, in the opinion of the investigator, might have interfered with the subject's participation in the study, posed an added risk for the subject, or confounded the assessment of the subject (e.g. severe cardiovascular, central nervous system or pulmonary disease).
13. Received BCV, CDV, ribavirin, or leflunomide within the previous 14 days.
14. Was receiving or was anticipated to need treatment with digoxin that could not have been withheld for the duration of BCV therapy.

Any exemptions to the protocol inclusion or exclusion criteria, as applicable, for subjects who developed probably or definitive AdV disease while participating in prescreening activities must have been discussed with and approved by the Chimerix medical monitor or designee before the subject was allowed to receive open-label BCV therapy.

Ages: 3 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Pheonix Children's Hospital, Phoenix, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Childrens hospital of LA, Los Angeles, California
  - CHOC Children's Hospital, Orange, California
  - University of California, San Francisco, San Francisco, California
  - Lucile Packard Childrens hopsital at Stanford, Stanford, California
  - The Children's Hospital-Denver, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Indiana University, Indianapolis, Indiana
  - LSU Health Sciences Center New Orleans Childrens Hospital, New Orleans, Louisiana
  - Harvard-Children's Hospital Boston, Boston, Massachusetts
  - Univeristy of Minnesota, Minneapolis, Minnesota
  - St. Louis Children's Hosptial, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Judes Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Baylor College of Medicine, Texas Childrens Hospital, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Methodist Hospital, San Antonio, Texas
  - Primary Children's Medical of Utah, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Result] Grimley MS, Chemaly RF, Englund JA, Kurtzberg J, Chittick G, Brundage TM, Bae A, Morrison ME, Prasad VK. Brincidofovir for Asymptomatic Adenovirus Viremia in Pediatric and Adult Allogeneic Hematopoietic Cell Transplant Recipients: A Randomized Placebo-Controlled Phase II Trial. Biol Blood Marrow Transplant. 2017 Mar;23(3):512-521. doi: 10.1016/j.bbmt.2016.12.621. Epub 2017 Jan 5. PMID 28063938
- [Derived] Tippin TK, Morrison ME, Brundage TM, Mommeja-Marin H. Brincidofovir Is Not a Substrate for the Human Organic Anion Transporter 1: A Mechanistic Explanation for the Lack of Nephrotoxicity Observed in Clinical Studies. Ther Drug Monit. 2016 Dec;38(6):777-786. doi: 10.1097/FTD.0000000000000353. PMID 27851688

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomized (blinded) subjects who considered treatment failures were offered open-label BCV therapy. These subjects followed the same schedule of assessments, beginning at Day 0 for up to 12 weeks followed by 4 weeks of post-treatment follow-up. Additionally, 4 subjects who had not been previously enrolled in the randomized (blinded) phase of the study were enrolled directly to the open-label arm.
Groups:
- Brincidofovir BIW: Randomized (Blinded) Phase
  * Adult subjects: 200 mg brincidofovir (BCV) administered as four 50 mg tablets taken orally twice weekly (BIW).
  * Pediatric subjects: 4 mg/kg BCV (not to exceed a total single dose of 200 mg) administered using a 10 mg/mL liquid formulation taken orally BIW (as 2 mg/kg).
- Brincidofovir QW: Randomized (Blinded) Phase
  * Adult subjects: 200 mg brincidofovir (BCV) administered as two 50 mg tablets taken orally once weekly (QW).
  * Pediatric subjects: 4 mg/kg BCV (not to exceed a total single dose of 200 mg) administered using a 10 mg/mL liquid formulation taken orally QW (as 4 mg/kg)
- Placebo: Randomized (Blinded) Phase
  * Adult subjects: Matching placebo tablets taken orally once weekly (QW; 2 tablets) or twice weekly (BIW; 4 tablets).
  * Pediatric subjects: Matching liquid placebo taken orally QW or BIW.
- Directly to Open-label: Subjects who were enrolled directly to open-label and had not been previously randomized (n=4) received 200 mg brincidofovir (BCV) administered as four 50 mg tablets taken orally twice weekly (BIW).
  This number does not include subjects who were previously randomized and moved to open-label (n=8), as they are represented in their previously randomized arm.
Period: Overall Study
Arm/Group | Brincidofovir BIW | Brincidofovir QW | Placebo | Directly to Open-label
Started | 14 | 16 | 18 | 4
Randomized to Open-label (The number of previously randomized subjects who were considered treatment failures were offered open-label BCV therapy.) | 3 | 4 | 5 | 0
Completed | 9 | 7 | 9 | 2
Not Completed | 5 | 9 | 9 | 2

BASELINE CHARACTERISTICS:
Population: Subjects in the Brincidofovir (BCV) BIW, BCV QW, and Placebo groups were randomized subjects who took at least 1 dose of study drug.
  Subjects in the BCV Open-Label group included 4 subjects who were not randomized and went directly into open-label, and 8 subjects from the BCV BIW and BCV QW groups. The baseline data represents the 4 subjects who were not previously randomized to the BCV BIW or BCV QW groups.
Groups:
- BCV BIW: Randomized (Blinded) Phase
  * Adult subjects: 200 mg brincidofovir (BCV) administered as four 50 mg tablets taken orally twice weekly (BIW).
  * Pediatric subjects: 4 mg/kg BCV (not to exceed a total single dose of 200 mg) administered using a 10 mg/mL liquid formulation taken orally BIW (as 2 mg/kg).
- BCV QW: Randomized (Blinded) Phase
  * Adult subjects: 200 mg brincidofovir (BCV) administered as four 50 mg tablets taken orally once weekly (QW).
  * Pediatric subjects: 4 mg/kg BCV (not to exceed a total single dose of 200 mg) administered using a 10 mg/mL liquid formulation taken orally QW (as 4 mg/kg).
- Placebo: Randomized (Blinded) Phase
  * Adult subjects: Matching placebo tablets taken orally once weekly (QW) or twice weekly (BIW).
  * Pediatric subjects: Matching liquid placebo taken orally QW or BIW.
- BCV Direct to Open-Label: Subjects who were enrolled directly to open-label and had not been previously randomized (n=4) received 200 mg brincidofovir (BCV) administered as four 50 mg tablets taken orally twice weekly (BIW).
  This number does not include subjects who were previously randomized and moved to open-label (n=8), as they are represented in their previously randomized arm.
- Total: Total of all reporting groups
Arm/Group | BCV BIW | BCV QW | Placebo | BCV Direct to Open-Label | Total
Number analyzed (Participants) | 14 | 16 | 18 | 4 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.6 (14.64) | 15.7 (20.67) | 13.8 (12.35) | 23.8 (21.55) | 14.8 (16.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 7 | 0 | 15
  Male | 9 | 13 | 11 | 4 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant AdV Infection
Description: The primary objective of this study was to evaluate the safety and efficacy of preemptive treatment with brincidofovir (BCV) versus placebo for the prevention of adenovirus (AdV) disease in recipients of hematopoietic stem cell transplantation (HCT) with asymptomatic AdV viremia.
  The outcome measure for the primary endpoint was treatment failure, a composite endpoint that consisted of the following:
  * Progression to probable AdV disease (other positive causes/agents have been ruled out and subject has disease-targeted organ-specific signs or symptoms) or definitive AdV disease (AdV detected in disease-targeted organ/system biopsy via antigen/immunohistochemistry, culture, and/or polymerase chain reaction and has at least 1 disease-targeted organ-specific sign or symptom); or
  * Increasing AdV viremia (defined as an increase from baseline in AdV viremia by ≥1 log10, confirmed on a second measurement, at least 1 week apart) and requiring discontinuation from blinded therapy.
Time Frame: 12 weeks
Population: Intent-to-Treat Population, defined as all randomized subjects who took at least 1 dose of study drug. Note that the subjects who were enrolled directly to open-label and not randomized are not included in this data.
Measure: Count of Participants; unit: Participants
Groups:
- BCV QW: Randomized (Blinded) Phase
  * Adult subjects: 200 mg brincidofovir (BCV) administered as two 50mg tablets taken orally once weekly (QW).
  * Pediatric subjects: 4 mg/kg BCV (not to exceed a total single dose of 200 mg) administered using a 10 mg/mL liquid formulation taken orally QW (as 4 mg/kg).
- Placebo: Randomized (Blinded) Phase
  * Adult subjects: Matching placebo tablets taken orally either once weekly (QW) or twice weekly (BIW).
  * Pediatric subjects: Matching liquid placebo taken orally either QW or BIW.
Arm/Group | BCV BIW | BCV QW | Placebo
Number analyzed (Participants) | 14 | 16 | 18
Participants | 3 | 6 | 6

ADVERSE EVENTS:
Description: Note that 8 subjects in the BCV open-label arm were previously randomized to 1 of the 3 blinded treatment arms: BCV BIW, BCV QW, or placebo. The adverse events reported for these subjects are presented according to what treatment arm they were under at the time the adverse event occurred.
Groups:
- BCV BIW: Randomized (Blinded) Phase
  * Adult subjects: 200 mg brincidofocir (BCV) administered as four 50mg tablets orally twice weekly (BIW).
  * Pediatric subjects: 4 mg/kg BCV (not to exceed a total single dose of 200mg) administered using a 10 mg/mL liquid formulation taken orally BIW (as 2 mg/kg).
- BCV QW: Randomized (Blinded) Phase
  * Adult subjects: 200 mg brincidofovir (BCV) administered as two 50mg tablets orally once weekly (QW).
  * Pediatric subjects: 4 mg/kg BCV (not to exceed a total single dose of 200mg) administered using a 10 mg/mL liquid formulation taken orally QW (as 4 mg/kg).
- Placebo: Randomized (Blinded) Phase
  * Adult subjects: Matching placebo tablets taken orally either once weekly (QW) or twice weekly (BIW).
  * Pediatric subjects: Matching liquid placebo taken orally QW or BIW.
- BCV Open-Label: Subjects who were enrolled directly to open-label and not randomized (n=4) and subjects who were previously randomized and moved to open-label (n=8) received 200 mg brincidofovir (BCV) administered as four 50 mg tablets taken orally twice weekly (BIW).
Arm/Group | BCV BIW | BCV QW | Placebo | BCV Open-Label
Serious Adverse Events (participants affected / at risk) | 6/14 | 7/16 | 6/18 | 8/12
Other Adverse Events (participants affected / at risk) | 13/14 | 14/16 | 16/18 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BCV BIW (N=14) | BCV QW (N=16) | Placebo (N=18) | BCV Open-Label (N=12)
BK virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Gingival abscess (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Acute graft versus host disease (Immune system disorders) | 2 | 2 | 1 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Metachromatic leukodystrophy (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BCV BIW (N=14) | BCV QW (N=16) | Placebo (N=18) | BCV Open-Label (N=12)
BK virus infection (Infections and infestations) | 3 | 3 | 2 | 2
Candidiasis (Infections and infestations) | 2 | 0 | 2 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 3 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 3
Klebsiella infection (Infections and infestations) | 0 | 0 | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Epstein-Barr viraemia (Infections and infestations) | 0 | 1 | 1 | 0
Human herpesvirus 6 infection (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Adenoviral upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1
Atypical mycobacterial pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Candida pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0
Encephalitic infection (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastrointestinal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia Klebsiella (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 0 | 0 | 1
Viral rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 6 | 5 | 6
Nausea (Gastrointestinal disorders) | 2 | 2 | 4 | 5
Vomiting (Gastrointestinal disorders) | 1 | 4 | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Caecitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lip blister (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 3 | 4 | 3
Fatigue (General disorders) | 1 | 3 | 0 | 0
Chills (General disorders) | 0 | 1 | 1 | 1
Implant site pain (General disorders) | 0 | 0 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 1 | 0
Medical device complication (General disorders) | 0 | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Fluid imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Food intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 4 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 1
Blood urea increased (Investigations) | 0 | 1 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 2 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 2
Weight increased (Investigations) | 0 | 0 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 0
Blood amylase increased (Investigations) | 1 | 0 | 1 | 0
Weight decreased (Investigations) | 2 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 1
Blood sodium increased (Investigations) | 0 | 0 | 0 | 1
Body temperature fluctuation (Investigations) | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1
Cardiac output decreased (Investigations) | 0 | 0 | 0 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 1
Fungal test positive (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0
Monocyte count decreased (Investigations) | 0 | 1 | 0 | 0
Polyomavirus test positive (Investigations) | 0 | 0 | 1 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 1 | 0 | 0
Acute graft versus host disease (Immune system disorders) | 7 | 4 | 3 | 5
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 1
Neurological symptom (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 3 | 2
Hypertension (Vascular disorders) | 0 | 1 | 0 | 2
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Refractoriness to platelet transfusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Gastrointestinal tube insertion (Surgical and medical procedures) | 0 | 0 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Gingival abscess (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metachromatic leukodystrophy (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 18 months after the end of the Study at all sites, if no publication of the overall multi-center results has been made, institutions are entitled to publish their locally obtained results, provided the Sponsor is given opportunity to review and comment. Institution publication may be delayed up to an additional 3 months to allow Sponsor to seek patent protection.